CLINICAL TRIAL: NCT07158710
Title: A Phase I, Open-label, Dose-escalation and Expansion Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HSK42360 in Pediatric Patients With BRAF V600-Mutant Malignant Brain Tumors
Brief Title: Phase I Study of HSK42360 in Malignant Brain Tumors With BRAF V600 Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK42360-103
Record Dates: First submitted 2025-08-06; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Malignant Brain Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ia: HSK42360 as monotherapy (Experimental): Phase 1a: dose escalation of HSK42360 as monotherapy at various dose levels
  Interventions: Drug: HSK42360
- Phase Ib: HSK42360 as monotherapy (Experimental): Phase 1b: dose expansion for HSK40118 as monotherapy at a dose determined during Phase 1a in patients with BRAF V600 recurrent mutation malignant brain tumors
  Interventions: Drug: HSK42360

INTERVENTIONS:
Drug: HSK42360 — Oral administration, QD/BID

SUMMARY:
This is a phase I, open-label, dose-escalation and expansion study to evaluate the safety, tolerability, PK of HSK42360 when given orally in pediatric patients with active BRAF V600 mutation recurrent malignant brain tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥6 and <18 years.
2. Karnofsky/Lansky Performance Status >60.
3. Life expectancy ≥ 3 months.
4. Patients with recurrent malignant brain tumors confirmed by histology or cytology, who have failed standard treatment (disease progression after treatment or intolerable treatment); patients who have previously received BRAF and/or MEK inhibitor therapy are allowed to be included in this study.
5. Positive BRAF V600 mutation result confirmed prior to the administration of HSK42360.
6. Patients will provide blood or tumor sample according to their own willingness.
7. Measurable disease by RANO criteria.
8. Patients with inactive CNS lesions, or patients treated with ≤5mg/day corticosteroid and without convulsion for ≥2 weeks.
9. Adequate hematologic, hepatic, and renal function.
10. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose.

Exclusion Criteria:

1. Patients with NF1 mutation.
2. malignant tumor within 2 years, with the exception of cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, or other tumors with low malignancy.
3. Uncontrollable pleural effusion, ascites, or pericardial effusion per protocol.
4. Treatment with any of the following:

   Prior treatment with anti-tumor drug within 4 weeks or approximately 5 × t1/2 prior to the first dose of HSK42360, whichever is shorter; Prior treatment with nitrosourea or mitomycin C within 6 weeks prior to the first dose of HSK42360; Prior treatment with palliative radiotherapy or anti-tumor herbs within 2 weeks prior to the first dose of HSK42360; Prior treatment with radiotherapy, electric field therapy, or other anti-tumor therapies within 4 weeks prior to the first dose of HSK42360.
5. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with the exception of alopecia, dermal toxicity, and other toxicity considering no safety risks by investigator.
6. Any disease which would preclude drug absorption, metabolism or pharmacokinetics, eg. active peptic ulcer or chronic gastroesophageal reflux disease.
7. Patient who have clinically significant or uncontrolled cardiac disease, include: QTc interval ≥ 450 msec; any clinically significant arrhythmia; left ventricular ejection fraction < 50%; myocardial infarction, unstable angina, or class III/IV cardiac failure by the NYHA that occurred within 6 months prior to the first dose of HSK42360.
8. Any thromboembolic events within 6 months prior to the first dose of HSK42360; any familial or aquired thrombophilia.
9. Any unstable systemic disease, eg. severe metabolic disease: liver cirrhosis, renal failure, or uremia.
10. Treatment with inhibitors/inducers for CYP3A4, or substrates of CYP3A4, CYP2C9, CYP2C8, OATP1B1, OATP1B3, OAT1, OAT3, P-gp or BCRP within 14 days or approximately 5 × t1/2 prior to the first dose of HSK42360, whichever is shorter.
11. Patient with cognitive dysfunction, or history of mental illness, other uncontrolled comorbidities, alcohol dependence, hormone dependence or drug abuse.
12. Autologous transplantation surgery within 3 months prior to the first dose of HSK42360; Allogeneic transplantation, or stem-cell Transplant surgery within 6 months prior to the first dose of HSK42360; Major surgery or significant traumatic injury occurring within 4 weeks prior to the first dose of HSK42360.
13. Patient with a history of immunodeficiency, including HIV positive, or other acquired/congenital immunodeficiency diseases.
14. Patient with severe retinal abnormalities and uveitis.
15. Patient with active hepatitis B or hepatitis C.
16. Allergic to any HSK42360 active constituent or ingredients.
17. Participate in other clinical trials within 4 weeks prior to the first dose of HSK42360.
18. Positive pregnancy test, or breastfeeding.
19. Any other circumstances that would, in the investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2029-05-23 (Estimated); Study Completion 2029-12-03 (Estimated)

PRIMARY OUTCOMES:
MTD | Up to approximately 52 months
  MTD determination: dose limiting toxicity (DLT) rate
DLTs | Up to approximately 52 months
  Incidence of dose-limiting toxicities (DLTs) at Cycle1
AEs | Up to approximately 52 months
  Rate and severity of adverse events of HSK42360 as monotherapy
RP2D | Up to approximately 52 months
  RP2D determination: DLT, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary safety and anticancer activity data
Karnofsky/Lansky Performance Scale | Up to approximately 52 months
  Change of the grade as a part of HSK43260 safety data

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 52 months
  ORR, defined as the proportion of patients who experience a best response of confirmed CR or PR according to RANO
Disease control rate (DCR) | Up to approximately 52 months
  DCR, defined as the proportion of patients who experience a best response of CR, PR, MR or stable disease (SD) according to RANO
Duration of response (DOR) | Up to approximately 52 months
  DOR, defined as the time from first documented response of CR, PR or MR to the date of first documented progressive disease or death due to any cause, whichever occurs first
Progression free survival (PFS) | Up to approximately 52 months
  PFS, defined as the time frocease or death due to any cause, whichever occurs first
Overall survival (OS) | Up to approximately 52 months
  OS, defined as the time from the first dose of HSK42360 until the date of death due to any cause
Area under the curve (AUC) | Circle 1 (28days)
maximum plasma concentration (Cmax) | Circle 1 (28days)
half-life (t1/2) | Circle 1 (28days)
Tmax(Time to maximum plasma concentration) | Circle 1 (28days)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Department of Neuro-oncology, Cancer Center, Beijing Tiantan Hospital, Capital Medical University,Beijing, China, Beijing, Beijing Municipality
  - The first affiliated hospital of fujian medical university, Fuzhou, Fujian
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Bethune Hospital of Jilin University, Changchun, Jilin
  - Fudan University Affiliated Huashan Hospital, Shanghai, Shanghai Municipality